CLINICAL TRIAL: NCT04758858
Title: Carbohydrates Under Target for Type 1 Diabetes Management
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not approved by REB
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Full professor, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUT-1
Record Dates: First submitted 2021-02-10; First posted 2021-02-17 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Pressure; Magnetic Resonance Spectroscopy; Hematologic Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VLCHF (Very Low CHO High Fat) Diet (Active Comparator): 10% of energy from CHO, 15% proteins, and 75% lipids
  Interventions: Other: Insulin treatment optimization with participant's usual diet; Device: Abbott's FreeStyle Libre; Other: Three-day food journal; Other: Medical visit; Other: Blood pressure measurements; Other: Anthropometric parameters measurements; Other: Indirect calorimetry test; Other: Well-being questionnaire; Other: Diet appreciation questionnaire; Device: Pedometer (PiezoRxD); Other: Hepatic imaging (MRI); Other: Glucagon efficiency test; Other: Body composition : Dual Energy X-ray absorptiometry (DEXA); Other: Blood tests; Other: Stool sample collections (optional); Other: Hypoglycemia journal; Other: Ketone journal; Other: Adherence to the diet (Keenoa)
- Low-CHO Diet (Active Comparator): 30% of energy from CHO, 15% proteins and 55% lipids
  Interventions: Other: Insulin treatment optimization with participant's usual diet; Device: Abbott's FreeStyle Libre; Other: Three-day food journal; Other: Medical visit; Other: Blood pressure measurements; Other: Anthropometric parameters measurements; Other: Indirect calorimetry test; Other: Well-being questionnaire; Other: Diet appreciation questionnaire; Device: Pedometer (PiezoRxD); Other: Hepatic imaging (MRI); Other: Glucagon efficiency test; Other: Body composition : Dual Energy X-ray absorptiometry (DEXA); Other: Blood tests; Other: Stool sample collections (optional); Other: Hypoglycemia journal; Other: Ketone journal; Other: Adherence to the diet (Keenoa)
- Control Diet (Placebo Comparator): 50% of energy from CHO, 15% proteins and 35% lipids
  Interventions: Other: Insulin treatment optimization with participant's usual diet; Device: Abbott's FreeStyle Libre; Other: Three-day food journal; Other: Medical visit; Other: Blood pressure measurements; Other: Anthropometric parameters measurements; Other: Indirect calorimetry test; Other: Well-being questionnaire; Other: Diet appreciation questionnaire; Device: Pedometer (PiezoRxD); Other: Hepatic imaging (MRI); Other: Glucagon efficiency test; Other: Body composition : Dual Energy X-ray absorptiometry (DEXA); Other: Blood tests; Other: Stool sample collections (optional); Other: Hypoglycemia journal; Other: Ketone journal; Other: Adherence to the diet (Keenoa)

INTERVENTIONS:
Other: Insulin treatment optimization with participant's usual diet — Two weeks before the intervention phase, insulin dose optimization and revision of participants' knowledge on carbohydrates counting, hypo- and hyperglycemia prevention and treatment will be done with a nurse and a dietitian under a physician's supervision. Once to twice a week, participants will be contacted to review if glucose values are in target.
Device: Abbott's FreeStyle Libre — During the whole trial, blood glucose will be assessed by intermittent scanning Continuous Glucose Monitors (isCGM; Abbott's Freestyle-Libre glucose sensor). Participants will be asked to record or download, in their Freestyle Libre reader or in their insulin pump, their insulin doses being injected each day.
Other: Three-day food journal — Two weeks before the intervention phase, participants will be asked to complete a 3-day food journal, using the Keenoa mobile application, with carbohydrates (CHO) content of food and blood glucose measures to optimize their insulin doses. Analysis of the food journal will allow us to quantify the participants' usual diet.
Other: Medical visit — During visit 1, a short medical interview will be done to establish if the subject is eligible to participate in the study. A list of current medications, presence of complications, as well as comorbidities associated with their diabetes will be collected in their medical file during the visit with the endocrinologist.
Other: Blood pressure measurements — Blood pressure (systolic and diastolic blood pressure) will be measured during all visits (visits 1 to 4).
Other: Anthropometric parameters measurements — Weight, height, BMI and waist circumference will be measured during all visits (visits 1 to 4).
Other: Indirect calorimetry test — Both resting metabolic rate and respiratory quotient will be measured after a 10-hour fast by indirect calorimetry. The test will be done twice, before (visit 2) and after (visit 4) the intervention phase.
Other: Well-being questionnaire — Participants will be asked to complete a well-being questionnaire (nausea, fatigue, etc) during visits 2, 3 and 4.
Other: Diet appreciation questionnaire — Participants will be asked to complete a diet appreciation (appetite, fullness, etc) questionnaire during visits 3 and 4.
Device: Pedometer (PiezoRxD) — Participants will be asked to wear a pedometer (PiezoRxD) that will record their steps every day during the whole trial. Also, they will have to install Piezo: Achieve the Guidelines!, a free mobile application, on their smartphone or tablet. It will connect to their pedometer via bluetooth and will help the research assistant track their data remotely
Other: Hepatic imaging (MRI) — Imaging of participants' liver will be done by MRI at the Centre Hospitalier de l'Université de Montréal (CHUM). The test will be done twice, before (visit 2) and after (visit 4) the intervention phase.
Other: Glucagon efficiency test — The glucagon efficiency test will be done twice, before (visit 2) and after (visit 4) the intervention phase. A subcutaneous insulin injection based on individual insulin correction factor will be given to induce hypoglycemia down to 3 mmol/L (based on plasma glucose). A subcutaneous injection of 300 µg of glucagon will be administered.
Other: Body composition : Dual Energy X-ray absorptiometry (DEXA) — Lean body mass and fat mass will be measured by Dual Energy X-ray absorptiometry (DEXA). The DEXA test will be done twice, before (visit 2) and after (visit 4) the intervention phase.
Other: Blood tests — Blood tests will be done to assess participants' diabetes control as well as to assess other biochemical markers (blood lipids as well as markers of inflammation and liver function). Blood will be collected and analyzed during all visits (visits 1 to 4).
Other: Stool sample collections (optional) — Participants will be asked to collect and immediately freeze their stool sample until it is given to the study team (for intestinal microbiota composition analysis). This will be done three times during the study, during phase 1, between week 1 and 6 of phase 2 and between week 6 and 12 of phase 2.
Other: Hypoglycemia journal — During the whole trial, participants will be asked to keep a log of their hypoglycemia episodes, which are defined by the need to consume CHO. They will be asked to note the time, symptoms (including time taken for disappearance after treatment), capillary glucose measurement and the amount of CHO consumed.
Other: Ketone journal — During the intervention phase, participants will be asked to measure their ß-hydroxybutarate level (mmol/L) with their Abbott's Freestyle-Libre scanner at least twice per week before breakfast. Participants will be asked to check their ketone bodies for sensor or capillary glucose levels exceeding 15 mmol/l, when their sensor indicates high without a specific glucose value and when they have symptoms of ketoacidosis (regardless of glucose reading).
Other: Adherence to the diet (Keenoa) — During the whole dietary intervention phase (phase 2), participants will confirm that they have followed their menus by taking before and after pictures of their meals every day and indicating the percentage of their meal consumed (25-50-75-100%) via the Keenoa mobile application.

SUMMARY:
Recently, there has been an increased interest in limiting carbohydrates (CHO) intakes for improving long-term health. Low CHO (<30% energy from CHO) and very low CHO high fat (VLCHF; 10% CHO, 75% Lipid) diets are being advocated among people living with diabetes given their almost immediate favorable impact on post-prandial blood glucose levels and on hemoglobin A1c that have been reported by users. Adoption of these diets are met with reluctance by healthcare professionals due to the lack of information on their safety. Concerns include the impact on hypoglycemia frequency and glucagon response to hypoglycemia, diabetic ketoacidosis, lipid profile, liver function insulin dose adjustments when adopting them in the context of type 1 diabetes (T1D). Through a series of interviews, people with diabetes following a VLCHF reported that the lack of support from HCPs often leads to hiding the fact that they have adopted a VLCHF diet. This is an important source of concern that can lead to additional safety issues.

The goal is to fill an important knowledge gap about the effectiveness, benefits and risks of low CHO and VLCHF diets for people with T1D. The primary objective is to compare the percentage of TIR of adults with T1D following a low-CHO diet or a VLCHF diet versus a control diet for 12 weeks. The secondary objectives are (1) to evaluate efficacy of glucagon in correcting hypoglycemia in the context of restricted carbohydrates intakes; (2) to evaluate changes in HbA1c at 12 weeks and glucose fluctuations and % of time in hypoglycemia at 6 weeks and 12 weeks of control diet, low-CHO diet or VLCHF diet; (3) to compare key cardiometabolic risk factors (body composition, blood lipids, blood pressure and liver inflammatory markers and function) at 6 weeks and 12 weeks of control diet, low-CHO diet or VLCHF diet; (4) to evaluate the effect of restrictive CHO diets (low-CHO and VLCHF) on the composition of the intestinal microbiota (optional).

ELIGIBILITY:
Inclusion Criteria:

* Men and women > 18 years old
* Duration of T1D > 12 months
* On intensive insulin therapy
* Own a smartphone or tablet to use two mobile applications for nutritional and physical activity tracking: Keenoa and Piezo: Achieve the Guidelines!

Exclusion Criteria:

* Already following a low-CHO diet (<30% CHO)
* Type 2 diabetes or other form of diabetes
* Known gastroparesis (clinical diagnosis)
* Advanced kidney disease (eGFR < 50 mL/min)
* Known significant liver disease (e.g. cirrhosis, active hepatitis, liver transplantation)
* Recent (<6 months) major cardiovascular event (e.g. myocardial infarction, cerebrovascular accident, major revascularization, etc.)
* Pregnancy (ongoing or planned in the next 6 months)
* Breastfeeding (ongoing)
* Recent severe hypoglycemia episodes (BG <2.8 mmol/L or assistance from a third party) or ketoacidosis (<6 weeks)
* Claustrophobia or presence of metal devices/implants in the body
* Recent (<6 weeks) or planned (next 6 months) modification in insulin treatment
* Recent (<6 weeks) or planned (next 6 months) modification in cardiometabolic drugs for blood pressure and/or lipids. These drugs must remain stable all along the trial
* Off label adjunct therapy with SGLT-2 inhibitors (Forxiga®, Invokana® or Jardiance®)
* Recent (<6 weeks) or planned (next 6 months) modification of adjunct therapy (Metformin, Glumetza®, Victoza®, Trulicity® and Ozempic®)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of time-in-target (range of 4-10 mmol/L) | From enrollment to end of study, total of 14 weeks
  Using continuous glucose monitoring (FreeStyle Libre)

SECONDARY OUTCOMES:
Time to resolve an induced hypoglycemia (>4 mmol/L) | After administration of subcutaneous insulin; At beginning (week 3) and end (week 14) of the diet intervention, each test lasts approximately 5 hours
  Glucagon efficiency test
Peak plasma glucose level two hours after glucagon administration | After administration of glucagon; At beginning (week 3) and end (week 14) of the diet intervention, each test lasts approximately 5 hours
  Glucagon efficiency test
Glycated hemoglobin (HbA1c) | During blood test : At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Average glycemic control
Fructosamine | During blood test : At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Average glycemic control
Fasting blood glucose | From beginning (week 3) to end (week 14) of diet intervention
  Blood glucose before meals
Post-prandial blood glucose | From beginning (week 3) to end (week 14) of diet intervention
  Blood glucose after meals
Coefficient of glucose variation (%) | From enrollment to end of study, total of 14 weeks
  Using continuous glucose monitoring (FreeStyle Libre)
Insulin daily dose | From enrollment to end of study, total of 14 weeks
  Using continuous glucose monitoring (FreeStyle Libre) or their insulin pump
Basal insulin doses | From enrollment to end of study, total of 14 weeks
  Using continuous glucose monitoring (FreeStyle Libre) or their insulin pump
Insulin-to-CHO ratio | From enrollment to end of study, total of 14 weeks
  Using continuous glucose monitoring (FreeStyle Libre) or their insulin pump
Percentage of time spent in hypoglycemia ranges < 4 mmol/L | From enrollment to end of study, total of 14 weeks
  Using continuous glucose monitoring (FreeStyle Libre)
Percentage of time spent in significant hypoglycemia ranges < 3 mmol/L | From enrollment to end of study, total of 14 weeks
  Using continuous glucose monitoring (FreeStyle Libre)
Weight (kg) | At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Weight and height will be combined to report BMI (kg/m^2)
Height (cm) | At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Weight and height will be combined to report BMI (kg/m^2)
Waist circumference (cm) | At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Calculated using the average of 3 measures
Total cholesterol | During blood test : At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Blood lipid profiles
HDL-cholesterol | During blood test : At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Blood lipid profiles
LDL-cholesterol | During blood test : At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Blood lipid profiles
Triglycerides | During blood test : At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Blood lipid profiles
Apo-B | During blood test : At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Blood lipid profiles
Apo-A1 | During blood test : At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Blood lipid profiles
Total lean mass (kg) | During DEXA-scan : At beginning (week 3) and end (week 14) of the diet intervention, each test lasts approximately 15 minutes
  Measured by DEXA (Dual-Energy X-ray Absorptiometry)
Total lean mass (%) | During DEXA-scan : At beginning (week 3) and end (week 14) of the diet intervention, each test lasts approximately 15 minutes
  Measured by DEXA (Dual-Energy X-ray Absorptiometry)
Truncal lean mass (kg) | During DEXA-scan : At beginning (week 3) and end (week 14) of the diet intervention, each test lasts approximately 15 minutes
  Measured by DEXA (Dual-Energy X-ray Absorptiometry)
Truncal lean mass (%) | During DEXA-scan : At beginning (week 3) and end (week 14) of the diet intervention, each test lasts approximately 15 minutes
  Measured by DEXA (Dual-Energy X-ray Absorptiometry)
Total fat mass (kg) | During DEXA-scan : At beginning (week 3) and end (week 14) of the diet intervention, each test lasts approximately 15 minutes
  Measured by DEXA (Dual-Energy X-ray Absorptiometry)
Total fat mass (%) | During DEXA-scan : At beginning (week 3) and end (week 14) of the diet intervention, each test lasts approximately 15 minutes
  Measured by DEXA (Dual-Energy X-ray Absorptiometry)
Truncal fat mass (kg) | During DEXA-scan : At beginning (week 3) and end (week 14) of the diet intervention, each test lasts approximately 15 minutes
  Measured by DEXA (Dual-Energy X-ray Absorptiometry)
Truncal fat mass (%) | During DEXA-scan : At beginning (week 3) and end (week 14) of the diet intervention, each test lasts approximately 15 minutes
  Measured by DEXA (Dual-Energy X-ray Absorptiometry)
Systolic blood pressure (mmHg) | At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Calculated using the average of 3 measures
Diastolic blood pressure (mmHg) | At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Calculated using the average of 3 measures
Aminotransferases | During blood test : At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Liver function
Alkaline phosphatase | During blood test : At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Liver function
Gamma-glutamyl transpeptidase | During blood test : At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Liver function
Bilirubin | During blood test : At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Liver function
Albumin | During blood test : At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Liver function
High sensitivity CRP | During blood test : At baseline (day 1), before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Liver function
Resting metabolic rate (kcal/day) | During indirect calorimetry test : At beginning (week 3) and end (week 14) of the diet intervention, each test lasts approximately 30 minutes
  Measured by indirect calorimetry
Respiratory quotient | During indirect calorimetry test : At beginning (week 3) and end (week 14) of the diet intervention, each test lasts approximately 30 minutes
  Measured by indirect calorimetry
Liver proton density fat fraction | During MRI : At beginning (week 3) and end (week 14) of the diet intervention, each test lasts approximately 30 minutes
  Hepatic fat imagery measured by MRI
Mean liver PDFF | During MRI : At beginning (week 3) and end (week 14) of the diet intervention, each test lasts approximately 30 minutes
  Hepatic fat imagery measured by MRI
Total liver volume | During MRI : At beginning (week 3) and end (week 14) of the diet intervention, each test lasts approximately 30 minutes
  Hepatic fat imagery measured by MRI
Total liver fat index | During MRI : At beginning (week 3) and end (week 14) of the diet intervention, each test lasts approximately 30 minutes
  Hepatic fat imagery measured by MRI
Well-being score | Before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  The World Health Organisation- Five Well-Being Index (WHO-5) : I have felt cheerful in good spirits, I have felt calm and relaxed, I have felt active and vigorous, I woke up feeling fresh and rested, My daily life has been filled with things that interest me. The raw score is calculated by totaling the figures of the five answers (0 = At no time to 5 = All of the time). The raw score ranges from 0 to 25, 0 representing worst possible and 25 representing best possible quality of life.
Visual Analog Score for fatigue (none to intolerable) | Before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Corresponding scores of questionnaire used to assess different quality of life aspects.
Visual Analog Score for nausea (none to intolerable) | Before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Corresponding scores of questionnaire used to assess different quality of life aspects.
Visual Analog Score for abdominal cramp/pain (none to intolerable) | Before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Corresponding scores of questionnaire used to assess different quality of life aspects.
Visual Analog Score for headache (none to intolerable) | Before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Corresponding scores of questionnaire used to assess different quality of life aspects.
Visual Analog Score for hunger (none to intolerable) | Before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Corresponding scores of questionnaire used to assess different quality of life aspects.
Visual Analog Score for diet satisfaction (not appreciated to very appreciated) | Before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Corresponding scores of questionnaire for diet appreciation.
Visual Analog Score for difficulty to follow the diet (no difficulty to extreme difficulty) | Before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Corresponding scores of questionnaire for diet appreciation.
Visual Analog Score for difficulty for meal preparation (no difficulty to extreme difficulty) | Before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Corresponding scores of questionnaire for diet appreciation.
Steps/day (physical activity) | From enrollment to end of study, total of 14 weeks
  Recorded with a pedometer (PiezoRxD) and mobile application
Number hypoglycemia episodes | From enrollment to end of study, total of 14 weeks
  Recorded by participants on hypoglycemia journal
Severity of hypoglycemia episodes (mild or severe) | From enrollment to end of study, total of 14 weeks
  Recorded by participants on hypoglycemia journal
Capillary ketone body levels | From beginning (week 3) to end (week 14) of diet intervention
  ß-hydroxybutarate level (mmol/L) measured using ketometer integrated in Abbott's Freestyle-Libre scanner
Alpha diversity (optional) | Before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Intestinal microbiota composition (optional)
Beta diversity (optional) | Before diet intervention (week 3), halfway the diet intervention (week 8) and at the end of the diet intervention (week 14)
  Intestinal microbiota composition (optional)
Daily caloric intake (kcal/day) | Three days during the first 2 weeks (3-day food journal) and from beginning (week 3) to end (week 14) of diet intervention
  Using Keenoa's mobile application
Lipids composition | Three days during the first 2 weeks (3-day food journal) and from beginning (week 3) to end (week 14) of diet intervention
  Using Keenoa's mobile application. Grams will be converted into percentage of energy.
Carbohydrates composition | Three days during the first 2 weeks (3-day food journal) and from beginning (week 3) to end (week 14) of diet intervention
  Using Keenoa's mobile application. Grams will be converted into percentage of energy.
Proteins composition | Three days during the first 2 weeks (3-day food journal) and from beginning (week 3) to end (week 14) of diet intervention
  Using Keenoa's mobile application. Grams will be converted into percentage of energy.
Self-reported symptoms | From enrollment to end of study, total of 14 weeks
  Descriptive symptoms reported by participants during follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada